CLINICAL TRIAL: NCT04195815
Title: A Pilot Study for Continuous Monitoring of Physical Activity Using Activity Armbands for 6 Months: Assessment of Feasibility and Comparison to Self-reported Questionnaires
Brief Title: Physical Activity Monitoring in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS)
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 28780
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2019-12

CONDITIONS: Chronic Fatigue Syndrome (CFS); Myalgic Encephalomyelitis (ME)
Keywords: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis; ME/CFS; Physical activity; Activity armband
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (serum, plasma, full blood) will be collected at baseline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will assess the feasibility of activity monitoring armbands for continuous measurement of physical activity level in ME/CFS patients, during 6 months follow-up. The main purpose is to assess if continuous measurement of activity level may be incorporated in outcome measures in future clinical interventional trials.

DETAILED DESCRIPTION:
The purpose is to assess feasibility of activity monitoring armbands for continuous measurement of physical activity level in patents with Myalgic Encephalopathy/ Chronic Fatigue Syndrome (ME/CFS), during 6 months follow-up.

The investigators will assess which physical activity parameters that best seem to reflect the participant's own perception of activity level, such as mean number of steps per 24 hours.

The investigators will assess the agreement between continuous activity measurements by activity armbands, and self-reported questionnaires for health-related quality of life (SF-36 ver.2) and for ME/CFS symptoms (DSQ-SF).

The investigators will assess the agreement between activity monitoring by armbands, and previously validated activity monitoring bracelets for 5-7 consecutive days, at baseline, at 3 months and at 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients wit ME/CFS according to Canadian Consensus Criteria (2003)
* ME/CFS disease duration at least 2 years
* Mild, Mild/moderate, Moderate, Moderate/Severe and Severe ME/CFS may be included
* Signed informed consent

Exclusion Criteria:

* Patients with fatigue, who do not meet the diagnostic "Canadian" criteria (2003) for ME/CFS
* ME/CFS disease duration < 24 months
* Patients where the diagnostic workup uncovers other pathology as possible cause of symptoms
* Serious endogenous depression
* Lack of ability to complete the study including follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 30 patients with ME/CFS according to Canadian Consensus Criteria (2003) with disease duration at least 2 years, of age 18-65 years
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Feasibility of activity monitoring armband to assess physical activity in ME/CFS patients | 6 months
  Feasibility of activity monitoring armbands to assess level of physical activity in ME/CFS patients, with comparison of activity data to self-reported questionnaires for quality of life (SF-36 ver.2) and for ME/CFS symptoms (DSQ-SF)

CONTACTS AND LOCATIONS:
Overall Officials: Olav Mella, MD, Prof, Study Director — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Rekeland IG, Sorland K, Bruland O, Risa K, Alme K, Dahl O, Tronstad KJ, Mella O, Fluge O. Activity monitoring and patient-reported outcome measures in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome patients. PLoS One. 2022 Sep 19;17(9):e0274472. doi: 10.1371/journal.pone.0274472. eCollection 2022. PMID 36121803